CLINICAL TRIAL: NCT02086851
Title: Impact of a Structured Parent Intervention on Weight Loss and Behavioral Change in Overweight Adolescents Enrolled in a Lifestyle Modification Program
Brief Title: Study of a Structured Parent Intervention on Adolescent Weight Loss Modification Program.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Children's Hospital Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM13833
Record Dates: First submitted 2014-02-07; First posted 2014-03-13 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Pediatric Obesity; Impact of Parent Intervention on Adolescent Weight Loss
Keywords: pediatric obesity; motivational interviewing; lifestyle intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Intervention plus Parent Motivational Interviewing (Experimental): Lifestyle intervention + Parent MI
  Interventions: Behavioral: Lifestyle Intervention; Behavioral: Parent Motivational Interviewing
- Lifestyle Intervention alone (Active Comparator): lifestyle intervention alone
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention
Behavioral: Parent Motivational Interviewing
  Arms: Lifestyle Intervention plus Parent Motivational Interviewing

SUMMARY:
The study will enroll 110 overweight and obese adolescents ages 11-16 in a lifestyle modification program focusing on dietary modification and exercise. Parents will be randomized into control and motivational interviewing-based intervention groups. The primary hypothesis is that adolescents whose parents are in the intervention group will have improved compliance, weight loss and health outcomes compared with adolescents whose parents do not receive the intervention.

DETAILED DESCRIPTION:
Adolescents will participate in a 6-month intensive lifestyle modification that includes a structured exercise program, nutrition education and dietary modification and behavioral support, followed by a 6-month maintenance phase with monthly booster sessions. Parents will be randomized to participate in 4 dedicated "pre-treatment" parent psychoeducational sessions vs. control (no psychoeducational sessions). The sessions will explore parents' feelings about participation in a weight management program, explore their reasons for wanting to make behavioral changes, and enhance motivation. All parents will participate in monthly parent support groups while their adolescents are participating in the intervention phase of the study. The 6-month adolescent intervention will include biweekly sessions with a registered dietitian for dietary education; biweekly interactive group discussion sessions on topics pertaining to motivation, strategies for changing health behaviors, setting and keeping goals and dealing with peer pressure; and exercise sessions three times a week with 30 minutes of cardiovascular exercise and 30 minutes of strength training each session. Comprehensive assessments, including nutrition, behavior and exercise assessments, laboratory work, body composition measurements and medical assessments will be conducted at baseline, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria: Age 11 - 16; BMI > 85th percentile; one parent or guardian committed to participate in protocol; -

Exclusion Criteria: Previous enrollment in IRB3354, IRB3008 or HM11113; Underlying genetic, neurological, endocrine or metabolic condition that preclude weight loss with conventional diet and exercise programs; Weight greater than 400 pounds, Pregnancy in female subjects; Inability to understand study instructions due to language barrier or mental disability; Primary residence outside a 30 mile radius of study location.

-

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2011-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in BMI z-scores | 12 weeks, 6 months and 12 months

SECONDARY OUTCOMES:
Changes in body composition | 12 weeks, 6 months and 1 year
Changes in BMI | 12 weeks, 6 months and 12 months
Changes in insulin sensitivity | 12 weeks, 6 months and 12 months
Changes in blood pressure | 12 weeks, 6 months and 12 months
Changes in serum lipids | 12 weeks, 6 months and 12 months
Changes in fitness measures | 12 weeks, 6 months and 12 months
Changes in ECG parameters | 12 weeks and 6 months
Changes I dietary intake | 12 weeks, 6 months and 12 months
Changes in quality of life scores | 12 weeks, 6 months and 12 months
Changes in BMI of participating parents | 12 weeks, 6 months and 12 months
Changes in body composition of participating parents | 12 weeks, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Edmond P Wickham, MD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- CHoR at VCU Healthy Lifestyles Center, Henrico, Virginia, United States